CLINICAL TRIAL: NCT05843526
Title: Influence of Implant Component Materials on Peri-implant Soft Tissue Host-response: A Randomized Clinical Trial.
Brief Title: Influence of Implant Component Materials on Peri-implant Soft Tissue Horst Response.
Acronym: PISTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B707201628072
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Dental Implants; Soft Tissue Inflammation; Immunohistochemistry; Dental Implants, Single-Tooth; Histology; Dental Implantation
Keywords: Dental implants; Soft Tissue Inflammation; Abutment materials; Immunohistochemistry; histometry; Peri implant tissues; dental material; Dental abutments; histology; peri implant tissue changes

STUDY DESIGN:
Intervention Model Description: The study included 69 implants divided into 3 groups. The 1st control group with titanium abutments, a second test group on dental resin (Optibond ™ FL, Kerr Dental) and a last test group on polyetheretherketone (PEEK).
Masking Description: Patient was allocated to a number. The collected samples were assigned to a reference number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Titanium abutment (Active Comparator): Titanium (Ti) grade 5 titanium abutment
  Interventions: Device: Experimental healing abutment
- Dental resin abutment (Experimental): Dental resin (Re) Optibond ™ FL, Kerr Dental abutment
  Interventions: Device: Experimental healing abutment
- Polyetheretherketone abutment (Experimental): Polyetheretherketone (PEEK) Polyetheretherketone abutment
  Interventions: Device: Experimental healing abutment

INTERVENTIONS:
Device: Experimental healing abutment — Implant placement (Straumann) Experimental abutment made of titanium, PEEK polyetheretherketone, resin was randomly assessed to the implant site.
  Abutment screw channel was filled with Teflon and closed with resin composite. Mouthwash based 0.2% chlorhexidine for 10 days and analgesics (ibuprofen 400 mg, up to 4/d) if necessary.
  After 8 weeks, harvesting of the soft tissues around experimental abutment with experimental abutment using a custom-made guide was placed on the experimental abutment

SUMMARY:
The aim of this study was to characterize the host-related response of peri-implant soft tissue induced by 3 different materials: titanium, resin and PEEK (polyetheretherketone) on man.

The primary endpoint is to asses the histological data available: Histological analyses are carried out with immunohistology (CD68, CD3, CD20, macrophages), non decalcified histology to appreciate the structure of the peri implant soft tissues (Sulcus depth, junctional epithelium, connective tissue adhesion).

Moreover: scanning electronic microscope (SEM) of the experimental abutment is performed to juge the cell adhesion on the abutment surface.

The secondary endpoint is to assess clinical data, radiological bone remodeling regarding the different material.

The hypothesis is that resin abutment lead to more inflammation than PEEK or titanium.

DETAILED DESCRIPTION:
The present study was designed as a randomized controlled trial. A total of 69 implants were placed and experimental abutments made of grade 5 titanium (Ti), dental resin (Optibond ™ FL, Kerr Dental)), polyetheretherketone (PEEK) were randomly allocated to each implant.

Study population: Patients needing tooth replacement in the posterior region (molars) are recruited from the Department of Periodontology and Oral and Implant Surgery of the University of Liege, Belgium.

Procedures

After a local anesthesia, implant procedure is carried out according to the recommendation of the manufacturer while considering the future position of the crown for a screw-retained restoration and the bone anatomy. Then, implants (Bone level or Bone level tapered, SLA active, Straumann Group, Basel, Switzerland) are placed with an insertion torque of at least 20 N/cm. The experimental abutment material is randomly allocated to the implant or two implants when it is possible: Titanium as a group control, PEEK (polyetheretherketone) or resin abutment.

The insertion is made at 15 N/cm and the access hole is obturated with teflon and Telio (Ivoclar vivadent, Schaan, Liechtenstein). A standardized parallel peri-apical radiograph is taken in order to record the baseline bone level. Each patient is instructed to rinse twice daily with an aqueous solution of 0,2% Chlorhexidine (Corsodyl®, GSK, Brentford, United Kingdom) and to avoid brushing of the area until the first recall 10-12 days later. Anti-inflammatories (Ibuprofen® 600 mg) as well as additional analgesics (Paracetamol® 500 mg) are recommended according to the patient's needs. Eight weeks after implantation, the buccal part of the abutment is marked with a drill, and a harvesting guide is placed on the experimental abutment. A punch device cut the soft tissue at 1mm from the abutment surface and both soft tissues and abutment are removed together. When the adherence between soft tissues and abutment is weak (soft tissues slide from the abutment), the abutment is analyzed alone on scanning electronic microscopy and the soft tissues alone are analyzed with immunohistochemistry. When adherence between the abutment and the soft tissues is sufficient, it goes to non decalcified histology. A screw retained abutment or a conventional healing abutment is placed after the harvesting procedure and the prosthetic rehabilitation is performed after 3 months of healing.

Follow-up evaluations and data recording are performed at inclusion visit (baseline), surgery and 8 weeks after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Needing implant therapy
* One or more missing teeth in the posterior area of either maxilla or mandible
* Good systemic health (ASA I/II)
* Full mouth plaque score (FMPI) lower than or equal to 25%
* The tooth at the implant site(s) had to be extracted or lost at least 12 weeks prior to implant placement
* 3 mm of keratinized mucosa in the bucco-lingual dimension with bone crest allowing at least a regular diameter implant (4.1 mm).

Exclusion Criteria:

* Autoimmune disease requiring medical treatment
* Medical conditions requiring prolonged use of steroids, use of bisphosphonates and denosumab intravenously or in oral use
* Pregnancy or breastfeeding women
* Alcoholism o chronical drug abuse
* Immunocompromised patients
* Uncontrolled diabetes
* Smokers (more than 5 cigs/day)
* Implant diameter under 4 mm (narrow implant)
* Infection (systemic or local)
* The site was excluded if it was previously treated with socket preservation techniques, presented untreated local inflammation, mucosal diseases or oral lesions, history of local irradiation therapy or persistent intraoral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Soft tissue inflammatory response | 8 weeks
  To evaluate the inflammatory response of the peri-implant soft tissue after 8 weeks in contact with the abutment material: Immunohistological analysis of the quantity of macrophages, neutrophils, B and T lymphocytes and blood vessels present in the different samples.
  It has been evaluated using markers: CD3, CD20, CD68, CD34 and counting of marked cells.
  Data are reported with semi quantitative scale.
Characterization of peri implant soft tissues | 8 weeks
  To determine the composition and the length of different parts of the peri implant soft tissues depending on subgingival abutment material (regarding the data of sulcus depth, junctional epithelium and connective tissue in mm) using non decalcified histology.

SECONDARY OUTCOMES:
dental plaque accumulation | 8 weeks
  To assess the amount of plaque present on the abutments with SEM analysis. semi quantitative analyses are performed on the abutment.
Peri-implant bone remodeling | 8 weeks
  Assessment of bone height changes using X-rays Radiographies are analyzed with software ImageJ and mesial and distal values of the bone remodeling (bone line to the implant shoulder) are collected in mm.
Soft tissue health changes assessed by Plaque Index | 8 weeks
  Assessment of plaque percentage
Soft tissue health changes assessed by Keratinized gingiva measure | 8 weeks
  Assessment of height of keratinized mucosa by probing in mm.
Soft tissue health changes assessed by soft tissues height | 8 weeks
  Assessment of height of soft tissue by probing in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Liège (CHU-Ulg), Liège, Belgium

IPD SHARING:
Plan to Share IPD: No